CLINICAL TRIAL: NCT02897453
Title: Retrospective Review With Prospective Surveillance of Safety and Efficacy in a Clinical Series of Spinal Tethering Patients
Brief Title: Safety and Efficacy Study of Spinal Tethering
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Zimmer Biomet (Industry)
Responsible Party: Sponsor
Other Study IDs: CSU2014-11S
Record Dates: First submitted 2016-07-14; First posted 2016-09-13 (Estimated); Last update posted 2020-08-20 (Actual); Status verified 2020-02

CONDITIONS: Adolescent Idiopathic Scoliosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- The Spinal Tethering System group: Patients with adolescent idiopathic scoliosis that have been implanted with the Spinal Tethering System in an anterior vertebral body tethering construct.
  Interventions: Device: The Spinal Tethering System

INTERVENTIONS:
Device: The Spinal Tethering System — An implant comprised of: vertebral body screws, vertebral body staples (washers), and a PET (polyethylene-terephthalate) cord.

SUMMARY:
This study is an opportunity to gather long term safety and efficacy information from patients who have had their scoliosis treated via anterior vertebral body tethering (VBT).

DETAILED DESCRIPTION:
Participants in this study will have already been implanted with a vertebral body tethering device. Patients will be recruited for prospective follow-up to enable systematic data capture from the point of study entry to their 18th birth year and skeletal maturity. Over the course of their follow-up clinical outcomes, patient reported outcomes, and radiographic outcomes will be tracked.

ELIGIBILITY:
Inclusion Criteria:

* Patients who assent/consent to participate in this study for prospective surveillance
* Patients at least 10 years old, inclusive, on the day of surgery
* Patients with idiopathic scoliosis
* Patient who has failed bracing (as defined by greater than 5° of progression and/or intolerance to brace wear)
* Patients who underwent an anterior vertebral body tethering procedure for treatment of scoliosis via thoracoscopic access or mini-thoracotomy
* Patients with a Lenke type 1 curve with lumbar modifier of A or B
* Patients whose pre-operative Cobb angle was ≥ 30° and ≤ 65°
* Patients whose pre-operative thoracic scoliometer reading is ≤ 20°
* Patients whose structural, thoracic curve bends out to ≤ 30° Cobb angle pre-operatively

  * Ideally supine bending film
  * Standing lateral bending film also acceptable
* Patients of Sanders stage ≤ 5 or Risser sign of ≤ 3 at the time of surgery
* Patients and parents that understand English

Exclusion Criteria:

* Patients with vertebral body staples at any level of their spine

  ---Specifically, vertebral body staples that span an intervertebral disc space and are implanted for fusionless correction of scoliosis
* Patients with any spine surgery prior to their VBT procedure
* Patients with any deformity correction surgery, on their Lenke 1 curve, after their VBT procedure
* With the exception of tether re-tensioning
* Patients with any vertebral bodies that were instrumented outside of a thoracoscopic or minithoracotomy approach in conjunction with their VBT procedure
* Patients that have an orthotic prescribed and used to correct their Lenke 1 curve any time after their VBT procedure but before the 2 year primary endpoint
* Patients who are pregnant
* Patients unwilling to return for prospective follow-up visit(s)
* Patients with major psychiatric disorders (as defined in DSM-5)
* Patients with a history of substance abuse (as defined in DSM-5)
* Patients who are wards of the court
* Patients who are in an active drug or device trial that is more than minimal risk and where their participation in the trial would confound the measurements of the present study
* Patients who are in a device trial for efficacy of a musculoskeletal device and where their participation in the trial would confound the measurements of the present study
* Patients who are less than 30 days out from completion from another clinical trial of more than minimal risk or for safety and efficacy
* Patients for whom the investigator deems unwilling/incapable of participating

Ages: 10 Years to 23 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Participants are individuals with idiopathic scoliosis who received surgical treatment utilizing a spinal tethering technique
Sampling Method: Non-Probability Sample
Enrollment: 56 (Actual)
Dates: Start 2016-07-06 (Actual); Primary Completion 2020-07-19 (Actual); Study Completion 2022-10 (Estimated)

PRIMARY OUTCOMES:
Cobb angle measurement of the patient's coronal deformity | 2 Years post Index Vertebral Body Tethering Surgery
  Coronal Cobb angle at 24 month follow up after vertebral body tethering
Quantification and timing of all adverse events | Up to 18 years of age or skeletal maturity is reached
  Patients will be followed until skeletal maturity or 18 years old; whichever is longer.

SECONDARY OUTCOMES:
Longitudinal changes in PedsQL (as available) | Yearly up to 2 years post index surgery. Biannually after 2 year post index surgery. Collected until patient is 18 or skeletally mature, whichever is longer.
  All prospective visits will capture the standard core scale of the PedsQL. This patient reported outcome is not standard of care therefore only prospective visits will capture the assessment.
Longitudinal changes in APPT (as available) | Yearly up to 2 years post index surgery. Biannually after 2 year post index surgery. Collected until patient is 18 or skeletally mature, whichever is longer.
  All prospective visits will capture the APPT (adolescent pediatric pain tool) score. This patient reported outcome is not standard of care therefore only prospective visits will capture the assessment.
Longitudinal changes in SRS-22 (as available) | Yearly up to 2 years post index surgery. Biannually after 2 year post index surgery. Collected until patient is 18 or skeletally mature, whichever is longer.
  All prospective visits will capture the SRS-22 (Scoliosis Research Society 22 item patient questionnaire) score. This patient reported outcome is not standard of care therefore only prospective visits will capture the assessment.
Longitudinal changes in thoracic kyphosis. | Yearly up to 2 years post index surgery. Biannually after 2 year post index surgery. Collected until patient is 18 or skeletally mature, whichever is longer.
Longitudinal changes in coronal balance | Yearly up to 2 years post index surgery. Biannually after 2 year post index surgery. Collected until patient is 18 or skeletally mature, whichever is longer.
Longitudinal changes in sagittal balance. | Yearly up to 2 years post index surgery. Biannually after 2 year post index surgery. Collected until patient is 18 or skeletally mature, whichever is longer.
Longitudinal changes in coronal Cobb angle. | Yearly up to 2 years post index surgery. Biannually after 2 year post index surgery. Collected until patient is 18 or skeletally mature, whichever is longer.
  In addition to the primary endpoint finding at 2 years post index surgery, this measure will assess durability of the coronal Cobb angle through skeletal maturity.
Longitudinal changes in thoracic spine height. | Yearly up to 2 years post index surgery. Biannually after 2 year post index surgery. Collected until patient is 18 or skeletally mature, whichever is longer.
  Capture of total vertical thoracic spine height at every post-surgical follow up until the patient is 18 years old or skeletally mature.

CONTACTS AND LOCATIONS:
Overall Officials: Amer Samdani, MD, Principal Investigator — Shriners Hospitals for Children - Philadelphia
Locations (1):
- Shriners Hospitals for Children, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: Undecided